CLINICAL TRIAL: NCT00459953
Title: Extended Cessation Treatment for Teen Smokers
Acronym: Nicoteens
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Joel D Killen, Principle Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA118035; R01CA118035 (NIH); NCT01330069 (obsolete NCT alias)
Record Dates: First submitted 2007-04-11; First posted 2007-04-13 (Estimated); Results first posted 2016-05-30 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-05

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Extended treatment (Experimental): extended cognitive behavioral treatment for smoking cessation; Participants receive an additional 9 sessions of cognitive behavior therapy
  Interventions: Drug: Extended treatment
- Control group (No Intervention): Monthly follow-up phone calls for assessment purposes and to control for potential therapeutic effects associated with continued contact

INTERVENTIONS:
Drug: Extended treatment — All participants receive an open label phase treatment that includes nicotine patch and cognitive behavior therapy for a period of 10 weeks. The extended treatment group received an additional 9 sessions of cognitive and behavioral skills training.
  Other Names: CBT; nicotine patch
  Arms: Extended treatment

SUMMARY:
This study is designed to test the efficacy of an extended smoking cessation program for teen smokers. We hypothesize that teen smokers randomized to extended treatment will have a higher abstinence rate at 52 week follow-up than teen smokers receiving only open label treatment.

DETAILED DESCRIPTION:
Adolescent smokers (aged 14-18; > 10 cigarettes/day) attending continuation high schools in the San Francisco-San Jose Bay Area will serve as the target population for this study. 280 smokers meeting eligibility criteria will be randomized. Our primary goal is to examine the effectiveness of a multi-factor extended treatment strategy in promoting longer-term smoking abstinence. All 280 smokers will receive 10 weeks of open label treatment consisting of nicotine patch therapy and group-based, intensive self-regulatory skills training (ST). Following open label treatment, half (n=140) will receive nine additional group-based ST sessions delivered over a 14 week period. Telephone counseling will also be provided in conjunction with an Interactive Voice Response system (IVR) that will allow early detection of smoking "slips" and rapid response by treatment staff. The other half (n=140) will not receive any additional therapy beyond that provided in the open label treatment phase. Abstinence and relapse will be assessed at the end of open label (10 weeks) and extended treatment (24 weeks) and at 52 weeks from the time of study entry. Our primary hypothesis is that smokers randomized to extended treatment will have a higher prolonged abstinence rate (PA) at 52 week follow-up than participants receiving only open label treatment. PA at 52 weeks will be the outcome measure used to evaluate the primary hypothesis and will be defined as a report of non-smoking following an initial 2-week grace period during which any smoking is not counted as a failure and an expired-air carbon monoxide level of <9PPM. Here, failure is defined as either seven consecutive days of smoking or smoking on at least one day on each of two consecutive weeks. Point prevalence abstinence will be examined as a secondary outcome and defined as no smoking, not even a puff, for seven consecutive days prior to assessment and an expired-air carbon monoxide level of <9PPM. With 150 participants per cell, we will have, in general, 80% power at a 2-tailed alpha of .05 to detect a difference in abstinence rates of at least 15% over a large range of success probabilities.

ELIGIBILITY:
Inclusion Criteria:

Age 14-18 at the beginning of the study

Smoking at least 10 cigarettes per day

At least one quit attempt in previous 6mos

Exclusion Criteria:

Current DSM-IV disorder (depression, panic disorder, social anxiety disorder and agoraphobia)

Current self report of daily or heavy use (more than three times per week) of any drugs (marijuana, alcohol, cocaine, opiates, stimulants, etc.)

Positive urine pregnancy test

Currently on bupropion (Wellbutrin, Wellbutrin SR, Zyban) or other antidepressants, MAOI's, antipsychotics, benzodiazepines

Currently on NRT

Currently receiving formal treatment for substance abuse problem, depression or anxiety

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 141 (Actual)
Dates: Start 2006-09; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel D Killen, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bailey SR, Harrison CT, Jeffery CJ, Ammerman S, Bryson SW, Killen DT, Robinson TN, Schatzberg AF, Killen JD. Withdrawal symptoms over time among adolescents in a smoking cessation intervention: do symptoms vary by level of nicotine dependence? Addict Behav. 2009 Dec;34(12):1017-22. doi: 10.1016/j.addbeh.2009.06.014. Epub 2009 Jul 5. PMID 19647373
- [Result] Bailey SR, Hagen SA, Jeffery CJ, Harrison CT, Ammerman S, Bryson SW, Killen DT, Robinson TN, Killen JD. A randomized clinical trial of the efficacy of extended smoking cessation treatment for adolescent smokers. Nicotine Tob Res. 2013 Oct;15(10):1655-62. doi: 10.1093/ntr/ntt017. Epub 2013 Mar 4. PMID 23460656

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The enrollment number in the protocol section (141) differs from the number of participants started in the participant flow module (143) because 2 of those originally enrolled were discovered to be living in the same household and assigned to different treatments. Thus, they were excluded from analyses.
Groups:
- Control Group: All participants receive an open label phase treatment that includes nicotine patch and cognitive behavior therapy for a period of 10 weeks. The control group received monthly follow-up phone calls for assessment purposes and to control for potential therapeutic effects associated with continued contact
Period: Overall Study
Arm/Group | Extended Treatment | Control Group
Started | 72 | 71
Completed | 71 | 70
Not Completed | 1 | 1
Not completed — not analyzed-household member in study | 1 | 1

BASELINE CHARACTERISTICS:
Population: Adolescent smokers were recruited from 10 continuation high schools in the San Francisco Bay Area over a period of 3 years. Recruitment was conducted on a nonrolling basis, with a new cohort participating each academic school year
Groups:
- Total: Total of all reporting groups
Arm/Group | Extended Treatment | Control Group | Total
Number analyzed (Participants) | 71 | 70 | 141
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 71 | 70 | 141
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 25 | 53
  Male | 43 | 45 | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 47 | 50 | 97
  Not Hispanic or Latino | 24 | 20 | 44
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 71 | 70 | 141

OUTCOME MEASURES:

1. Primary Outcome: Point Prevalence Abstinence
Description: Point prevalence abstinence is defined as a report of nonsmoking (not even a puff) for 7 consecutive days prior to assessment and an expired-air carbon monoxide level below 9 parts per million (ppm)
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Extended Treatment | Control Group
Number analyzed (Participants) | 71 | 70
participants | 15 | 5

ADVERSE EVENTS:
Arm/Group | Extended Treatment | Control Group
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/71
Other Adverse Events (participants affected / at risk) | 22/71 | 22/70
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extended Treatment (N=71) | Control Group (N=70)
Nausea (Gastrointestinal disorders) | 12 (12) | 12 (12)
Lightheaded (General disorders) | 11 (11) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No